CLINICAL TRIAL: NCT02529761
Title: Transarterial Chemoembolization (TACE) With or Without Sorafenib in Intermediate Stage Hepatocellular Carcinoma: a Multicenter Prospective Nonrandomized Study
Brief Title: TACE With or Without Sorafenib in Intermediate Stage Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Director, Air Force Military Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-T 002
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; sorafenib; TACE; overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib combined with TACE (Experimental): 220 subjects in this study group will receive the treatment of sorafenib combined with conventional TACE.
  Interventions: Drug: Sorafenib; Procedure: TACE
- TACE monotherapy (Active Comparator): 110 subjects in this study group will receive the treatment of conventional TACE monotherapy.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: Sorafenib — Sorafenib will be supplied as 200 mg tablets. All subjects will take two tablets of sorafenib (200 mg tablets) twice daily (each morning and evening).
  Other Names: •Bay 43-9006, Sorafenib (Nexavar®)
  Arms: Sorafenib combined with TACE
Procedure: TACE — The first treatment of TACE should be completed within 3-7 days after the administration of sorafenib started. In all cases, TACE consists of an injection containing a mixture of chemotherapeutic agents and lipiodol followed by embolization with polyvinyl alcohol (PVA) particles until complete stasis was achieved in the tumor-feeding vessels.Tumor-feeding vessels should be selected/superselected whenever possible. TACE will be repeated "on demand" depending on the radiological response.
  Other Names: conventional transarterial chemeombolization

SUMMARY:
This multicenter prospective nonrandomized study is to evaluate the efficacy of TACE combined with sorafenib compared with TACE monotherapy in term of overall survival in intermediate-stage HCC.

DETAILED DESCRIPTION:
Sorafenib, a multikinase inhibitor, has been successfully applied for solid tumors such as renal cancer and HCC.

According to the Barcelona Clinic Liver Cancer (BCLC) staging classification, transarterial chemoembolization (TACE) has been recommended as a first line-therapy for patients at intermediate stage - BCLC B class (multinodular asymptomatic tumors without an invasive pattern).

Because sorafenib may improve the efficacy of locoregional therapy by decreasing post-TACE angiogenesis, sorafenib in combination with TACE has attracted considerable attention as a promising therapy

ELIGIBILITY:
Inclusion Criteria:

1. Prior informed consent
2. Intermediate stage HCC/ BCLC B stage
3. Confirmed Diagnosis of HCC:

   1. Cirrhotic subjects: Clinical diagnosis by AASLD criteria. HCC can be defined in cirrhotic subjects by one imaging technique (CT scan, MRI, or second generation contrast ultrasound) showing a nodule larger than 2 cm with contrast uptake in the arterial phase and washout in venous or late phases or two imaging techniques showing this radiological behavior for nodules of 1-2 cm in diameter. Cytohistological confirmation is required for subjects who do not fulfill these eligibility criteria.
   2. Non-cirrhotic subjects: For subjects without cirrhosis, histological or cytological confirmation is mandatory. Documentation of original biopsy for diagnosis is acceptable
4. Child Pugh class A/B(7) class without ascites or hepatic encephalopathy
5. ECOG Performance Status of 0-1
6. At least one uni-dimensional lesion measurable by CT-scan or MRI according to the RECIST 1.1, mRECIST and EASL criteria, respectively.

   1. Single lesion>5cm
   2. 2-3 lesions, at least one lesion>3cm; if more than 4 lesions, no limitation of the tumor size, but the sum of size of all tumor lesions should be less than 50% of liver parenchyma.
7. Male or female subject ≥ 18 years of age
8. Ability to swallow oral medications
9. Life expectancy of at least 12 weeks
10. Pregnancy test negative within 14 days before treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial
11. Adequate bone marrow, liver and renal functions as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to randomization:

    1. Hemoglobin > 9.0 g/dl
    2. Absolute neutrophil count (ANC) >1,500/mm3
    3. Platelet count ≥50x109/L
    4. ALB ≥28g/L
    5. Total bilirubin < 2 mg/dL
    6. ALT and AST < 5 x upper limit of normal
    7. BUN and creatinine < 1.5 x upper limit of normal
    8. INR < 1.7, or PT < 4 seconds above control

Exclusion Criteria:

1. Diffuse HCC or tumor size ≥50% of liver parenchyma
2. Vascular invasion
3. Presence of extrahepatic metastasis
4. Poor blood supply for the liver tumor lesions; poor blood supply refers that the tumor lesions fail to show obvious contrast uptake in the arterial phase and washout in venous or late phases by CT scan or MRI
5. Any contraindications for hepatic embolization procedures:

   1. Known hepatofugal blood flow
   2. Known porto-systemic shunt
   3. Renal failure / insufficiency requiring hemo-or peritoneal dialysis
6. Target lesions having previously been treated with local therapy such as resection of HCC, radiofrequency ablation (RFA), percutaneous ethanol injection (PEI)
7. Investigational drugs or other molecular target drugs ongoing or completed < 4 weeks prior to the baseline scan
8. Prior transarterial embolization or anti-tumor systemic chemotherapy
9. Any ≥ CTC AE grade 2 acute toxic effects of any prior local treatment
10. Patients with untreated varices or active bleeding
11. History of cardiac disease:

    1. Congestive heart failure >New York Heart Association (NYHA) class 2
    2. Uncontrolled hypertension
12. Known history of HIV infection
13. Active clinically serious infections (> grade 2 NCI-CTCAE Version 4.0), except for HBV and HCV infection
14. Clinically significant gastrointestinal bleeding within 4 weeks prior to start of study drug
15. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months prior to the first dose of study drug
16. Previous or concurrent cancer that is distinct in primary site or histology from HCC. Any cancer curatively treated >3 years prior to entry is permitted
17. Any contraindication for sorafenib or doxorubicin administration
18. Pregnant or breast-feeding subjects
19. Any disease which could affect the evaluation of the study drug: unstable angina, active CAD, uncontrolled arrhythmias, and myocardial infarction
20. Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study
21. Major surgery within 4 weeks prior to start of study drug (e.g. thoracolaparotomy is not allowed, but noninvasive surgery, e.g. biopsy, is allowed)
22. Autologous bone marrow transplant or stem cell rescue within 1 year prior to start of study drug
23. History of organ allograft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2015-08; Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | The last patient has been on study for 1.5 year
  Overall survival analysis is measured from the treatment start until death occurred from any cause

SECONDARY OUTCOMES:
Time to progression | The time to progression will be assessed at the end of the study, up to 3 years
  The time to progression is measured from the treatment start to the radiologically confirmed progression
Tumor response | Tumor response will be assessed at week 4 and week 8 after initiation of treatment and thereafter every 8 weeks (±7 days), up to 3 years
  Tumor response will be evaluated according to RECIST, mRECIST and EASL criteria, respectively. Tumor response will be presented in the terms of complete response, partial response, stable disease and progression disease
Adverse events | The adverse events will be assessed every 4 weeks, up to 3 years
  The terms and grade of adverse events will be presented according to the Common Terminology Criteria for Adverse Events(CTCAE:version 4.0)
Prognostic factor | The analysis will be perfomed when the last patient has been on study for 1.5 year
  The Cox proportional model will be used to assess the prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, MD, Principal Investigator — Xijing Hospital of Digestive Disease, Fourth Military Medical University
Locations (1):
- Xijing Hospital of digestive disease, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Result] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Result] Zhao Y, Wang WJ, Guan S, Li HL, Xu RC, Wu JB, Liu JS, Li HP, Bai W, Yin ZX, Fan DM, Zhang ZL, Han GH. Sorafenib combined with transarterial chemoembolization for the treatment of advanced hepatocellular carcinoma: a large-scale multicenter study of 222 patients. Ann Oncol. 2013 Jul;24(7):1786-1792. doi: 10.1093/annonc/mdt072. Epub 2013 Mar 18. PMID 23508822